CLINICAL TRIAL: NCT06751043
Title: FEEDS Trial - Fasting Preprocedurally in Enteral Nutrition: Evaluation of Divergent Approaches in Secure Airway
Brief Title: Preoperative Fasting vs. Not Fasting in Critically Ill Patients
Acronym: FEEDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Alexander Nagrebetsky, MD MSc, Anesthesia Attending, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024P003035; BPS-2023C1-31273 (Other Grant/Funding Number: PCORI - Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; Surgical Procedure, Unspecified; Pulmonary Aspiration; Fasting
Keywords: pulmonary aspiration; enteral nutrition; tube feeding; preoperative fasting; perioperative medicine; surgery in critically ill; procedures in critically ill; nutrition in critical illness; perioperative safety; preoperative management; preoperative fasting in secure airway; anesthesia in critically ill
MeSH Terms: conditions — Critical Illness; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Phase III pragmatic multicenter parallel-group randomized controlled non-inferiority trial with patient-level randomization and assessor blinding. If non-inferiority is demonstrated, we will perform a pre-specified superiority test.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (Active Comparator): Patients randomized to the Fasting arm will have tube feeding stopped at least 8 hours before the scheduled surgery or procedure time.
  Interventions: Other: Fasting
- Not Fasting (Active Comparator): Patients randomized to the Not Fasting arm will have tube feeding continued until transfer to the operating room/procedure area.
  Interventions: Other: Not fasting

INTERVENTIONS:
Other: Fasting — Process: Fasting pre-procedure
  Tube feeding will be stopped at least 8 hours before the patient's scheduled surgery or procedure time.
  Arms: Fasting
Other: Not fasting — Process: Not fasting pre-procedure
  Tube feeding will be continued until patient transfer to the operating room/procedure area.
  Arms: Not Fasting

SUMMARY:
The goal of this clinical trial is to learn if fasting or not fasting before a procedure has an effect on recovery in those who are critically ill. The main questions it aims to answer for patients on a breathing machine who are receiving tube feeding are:

* Does the risk of lung complications and death differ between those who are not fasting, which may have a higher chance of allowing tube feeding to enter the lungs, and fasting, which temporarily stops nutrition before a procedure?
* Is there a difference in recovery times, hospital stays, infection rates, need for organ support, safety, and nutrition for those who either fast or do not fast before a procedure?
* What is the relationship between nutrition and clinical outcomes?

Researchers will compare not fasting and fasting to see if it has an effect on recovery.

Participants will:

* Be assigned by chance (like a coin toss) to one of two groups. One group (fasting group) will have their tube feeding stopped at least 8 hours before their procedure. The other group (not fasting group) will have their tube feeding stopped right before their procedure.
* Be monitored via medical record for amount of protein and calories received, and any complications related to fasting/not fasting.
* Receive a phone call from the study team about 3 months after they enter the study to see how they are doing and complete a questionnaire.

'

DETAILED DESCRIPTION:
Patient Population: Critically ill patients in the ICU who are: mechanically ventilated, receiving tube feeding (enteral nutrition), with a planned surgery or procedure. Up to 1072 subjects will be enrolled.

Phase III pragmatic multicenter parallel-group randomized controlled non-inferiority trial with patient-level randomization and assessor blinding.

Enrollment Period: Approximately two years.

Aims:

* Aim 1: To compare the risk of pulmonary complications and mortality from: (1) perioperative pulmonary aspiration6,33,34 due to not fasting vs. (2) systemic effects of nutritional loss18-24 due to preoperative fasting. We will quantify the risk of pulmonary complications and mortality as the number of postoperative days alive and free from mechanical ventilation (DAFV)35,36 in the target population of critically ill patients with a secure airway who undergo interventional procedures.
* Aim 2: To compare length of ICU and hospital stay, discharge to home, need for organ support, infectious complications, safety outcomes, and nutritional outcomes in tube-fed mechanically ventilated patients with a secure airway who are fasted vs. not fasted prior to procedure.
* Aim 3: To define the relationship between perioperative fasting duration, calorie/protein delivery, and clinical outcomes in mechanically ventilated patients who receive tube feeding.

Study participants will be randomized with a 1:1 allocation ratio to one of the following preprocedural interventions:

1. Fasting - stopping tube feeding at least 8 hours prior to the scheduled procedure time;
2. Not fasting - tube feeding until call for transfer to the procedure area.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Age ≥ 18
2. Current admission to ICU*
3. Secure airway** with no plans for its removal prior to procedure
4. Current non-trophic (> 10 mL/hr) tube (enteral) feeding*** with no plans to discontinue prior to procedure for reasons other than preoperative fasting
5. Planned eligible procedure (Examples are listed in Appendix C) with anesthesia care or nursing sedation. Eligible procedures are defined as non-emergent diagnostic or therapeutic interventions that:

   * Do NOT have a well-established practice of preoperative fasting. (For example, bedside placement of a vascular catheter [arterial, central venous, peripheral venous] by the ICU team is NOT eligible for this trial since it has a widely established practice of no preoperative fasting and is not generally scheduled for a specific time.)
   * Do NOT require fasting for preoperative gastrointestinal tract preparation
   * Do NOT require removal/replacement of the endotracheal or tracheostomy tube
   * Do NOT require prone or Trendelenburg (head-down) positioning.
   * Typically require procedural sedation or anesthesia care.
   * Generally, are scheduled for a specific time (although this time can change, or procedure may be cancelled).
   * Are performed in the operating room, non-operating room procedural areas, or at the patient's bedside.

     * All ICU types are eligible: surgical, medical, cardiac, neurological, trauma, mixed etc.

       * Secure airway is defined as a cuffed endotracheal tube or a cuffed tracheostomy tube.

         * Patients with all types of feeding tubes are eligible, regardless of tube insertion site (nasal, oral, surgically implanted) and tube tip location (pre- and post-pyloric) †As determined by the enrolling physician-investigator

Exclusion Criteria

1. Inability to obtain informed consent
2. Inability to enroll and randomize > 8 hours prior to planned procedure time
3. Inability to deliver trial interventions
4. Expected survival < 48 hours as determined by the enrolling physician-investigator
5. Critically ill burn patient
6. Emergency procedure
7. a. Gastrointestinal tract procedure that requires fasting based on surgical indications or b. airway/lung procedure that requires removal of endotracheal or tracheostomy tube
8. Plan for prone or Trendelenburg (head down) positioning during most of the procedure
9. Major impairment of gastrointestinal motility or major structural disease of the gastrointestinal tract (e.g., severe gastroparesis, bowel obstruction, severe ileus, severely compromised lower esophageal sphincter, active gastrointestinal bleeding)
10. Plan for postoperative extubation in the procedure area
11. Prisoner
12. Pregnant woman, woman of childbearing potential without a documented negative urine or serum pregnancy test during the current hospitalization, or woman who is breast feeding
13. Refusal to enroll patient by treating physician
14. Extracorporeal Membrane Oxygenation (ECMO) at the time of potential enrollment, except patients scheduled for ECMO decannulation as the study procedure and patients expected to be off of ECMO at the time of study procedure.
15. Chronic mechanical ventilation at pre-admission level of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Days alive and free from mechanical ventilation on postoperative day 28. | Post-operative day 28
  Defined as the days alive and free of organ support (dialysis, assisted ventilation, and vasopressors) to day 28. Participants will need to be free of all three components (assisted ventilation, vasopressors, new renal replacement therapy) to qualify for a day alive and free from organ failures. Patients on chronic dialysis will not be scored for the new renal failure free component of this outcome.

SECONDARY OUTCOMES:
Postoperative mortality | Post-operative day 28
  Death from any cause at any location, including deaths after withdrawal of care.
Ventilator-free days in survivors | Post-operative day 28
  28 minus last post-operative day of mechanical ventilation assessed only in survivors at post-operative day 28. Non-survivors are excluded
All-cause, all-location mortality | Post-operative day 90
  Death from any cause at any location, including deaths after withdrawal of care.
Length of ICU stay | Post-operative day 90
  90 minus the last post-operative day of ICU admission.
Length of hospital stay | Post-operative day 90
  90 minus the last post-operative day of hospital/facility admission.
Days alive and without life support54 Days alive and without life support | Post-operative day 90
  90 minus the last post-operative day of mechanical ventilation, renal replacement therapy, or circulatory support (ECMO, vasopressor or inotrope), whichever is used last.
Proportion of patients alive and at home | Post-operative day 90
  Proportion of patients who are alive and at home or at pre-index hospitalization level of care.
Health-related quality of life | Post-operative day 90
  Short-Form 20
New surgical site infection | Post-operative day 90
  Documentation of superficial incisional or organ/space infection after index procedure in routine medical records
New bacteremia | Post-operative day 90
  Bacteremia in patients without pre-study intervention evidence of bacteremia during the same hospital admission.
Perioperative pulmonary aspiration | Time of procedure start +/- 24 hours
  Periprocedural pulmonary aspiration of gastric contents documented in routine medical records.
Perioperative Hyperglycemia | Time of procedure start +/- 24 hours
  Routinely collected blood glucose of > 180 mg/dL on at least one measurement.
Perioperative hypoglycemia | Time of procedure start +/- 24 hours
  At least one episode of routinely collected blood glucose of 41 to 70 mg/dL (moderate hypoglycemia) or ≤ 40 mg/dL (severe hypoglycemia).
Preoperative fasting duration | Time of procedure start - 72 hours
  Time from last routinely documented non-trophic (> 10 mL/hr) tube feeding to procedure start.
Postoperative fasting duration | Time of procedure start + 72 hours
  Time from procedure end to the first routinely documented non-trophic (>10 mL/hr) tube feeding volume/rate.
Perioperative fasting duration | Time of procedure start +/- 72 hours
  Duration of preoperative plus postoperative fasting.
Preoperative calories delivered | Time of procedure - 72 and -24 hours
  Total number of calories delivered via tube feeding within 24 and 72 hours prior to procedure.
Postoperative calories delivered | Time of procedure + 72 and + 24 hours
  Total number of calories delivered via tube feeding within 24 and 72 hours after the procedure.
Perioperative calories delivered | Time of procedure +/- 72 and +/- 24 hours
  Total number of calories delivered via tube feeding within 24 and 72 hours of the procedure.
Preoperative protein delivered | Time of procedure - 72 and -24 hours
  Total amount of protein delivered via tube feeding within 24 and 72 hours prior to procedure.
Postoperative protein delivered | Time of procedure + 72 and + 24 hours
  Total amount of protein delivered via tube feeding within 24 and 72 hours after the procedure.
Perioperative protein delivered | Time of procedure +/- 72 and +/- 24 hours
  Total amount of protein delivered via tube feeding within 24 and 72 hours of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Nagrebetsky, MD, MSC, Principal Investigator — Massachusetts General Hospital
Locations (19):
- United States (19):
  - Stanford Medical Center, Palo Alto, California
  - UCSF Medical Center Parnassus, San Francisco, California
  - University of Colorado Medical Center, Aurora, Colorado
  - University of Miami Hospital, Miami, Florida
  - McGaw Medical Center of Northwestern, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Columbia University Irvine Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Medical Branch, Galveston, Texas
  - UT Health Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study sites of this trial will share deidentified data through eCRF with the Statistical and Data Coordinating Center. The shared data will include patient baseline characteristics (clinical and demographic), data on trial interventions, and outcome data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion of the study, the final cleaned and locked data set will be deidentified per the HIPAA Privacy Rule (45 C.F.R. § 164.514(b)). The deidentified Full Data Package will be deposited in the Patient-Centered Outcomes Data Repository (PCODR) at the Inter-university Consortium for Political and Social Research (ICPSR) at the University of Michigan.
Access Criteria: Access to the data will be based on the regulations of the Patient-Centered Outcomes Data Repository (PCODR) at the Inter-university Consortium for Political and Social Research (ICPSR) at the University of Michigan.